CLINICAL TRIAL: NCT00790036
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Phase III Study of RAD001 Adjuvant Therapy in Poor Risk Patients With Diffuse Large B-Cell Lymphoma (DLBCL) of RAD001 Versus Matching Placebo After Patients Have Achieved Complete Response With First-line Rituximab-chemotherapy
Brief Title: Phase III Study of RAD001 Adjuvant Therapy in Poor Risk Patients With Diffuse Large B-Cell Lymphoma (DLBCL) of RAD001 Versus Matching Placebo After Patients Have Achieved Complete Response With First-line Rituximab-chemotherapy
Acronym: PILLAR2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRAD001N2301; 2008-000498-40 (EudraCT Number)
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse large B cell lymphoma; DLBCL; poor risk; R-IPI 3-5; adjuvant therapy; after R-CHOP or R-EPOCH; after R-CHOP; B-cell lymphoma; lymphoma; b cells; blood cancer; lymph nodes; Hodgkin's; non-Hodgkin
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Lymphoma; Hematologic Neoplasms | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Everolimus (Experimental): Participants who received Everolimus 10 mg (two 5 mg tablets), daily for 12 months
  Interventions: Drug: Everolimus
- Placebo (Placebo Comparator): Participants who received Everolimus placebo 10 mg (two 5 mg tablets), daily for 12 months
  Interventions: Drug: Everolimus Placebo

INTERVENTIONS:
Drug: Everolimus — Everolimus was formulated as tablets of 5 mg strength, blister-packed under aluminum foil in units of 10 tablets.
  Other Names: RAD001
  Arms: Everolimus
Drug: Everolimus Placebo — Everolimus placebo was formulated as tablets of 5 mg strength, blister-packed under aluminum foil in units of 10 tablets.
  Arms: Placebo

SUMMARY:
Phase III study of RAD001 adjuvant therapy in poor risk patients with Diffuse Large B-Cell Lymphoma (DLBCL) of RAD001 versus matching placebo after patients had achieved complete response with first-line rituximab-chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients with previous histologically confirmed Stage III-IV (or Stage II bulky disease, defined as any tumor mass more than 10 cm in longest diameter), at time of original diagnosis, diffuse large B cell lymphoma (pathology report based on original tumor tissue/lymph node is acceptable for meeting inclusion criteria, but tumor tissue (slides/block) must be available to be sent for central pathology to confirm diagnosis).
2. Patients defined as poor risk with IPI of 3, 4, or 5 at time of original diagnosis.
3. Patients age ≥ 18 years old.
4. Patients must have achieved complete remission (CR) based on the revised IWRC (Cheson et al 2007) following first line R-chemotherapy treatment. Radiation therapy (RT) during or after R-chemotherapy is acceptable provided: 1) it ends 4 weeks prior to start of study drug and, 2) in case of consolidation RT targeted at initial bulky tumor mass, administered after R-chemotherapy, patient is already in CR before initiating RT. Complete remission from R-chemotherapy must be confirmed by clinical and radiologic evaluation along with bone marrow confirmation (if bone marrow was involved by lymphoma before the R-chemotherapy treatment). Local pathology report on the bone marrow biopsy is acceptable. If bone marrow was not involved by lymphoma before R-chemotherapy treatment, then bone marrow confirmation after R-chemotherapy is not required.
5. Patients who received a minimum 5 cycles of R-chemotherapy treatment and maximum 8 cycles of R-chemotherapy treatment. Any variation of CHOP (R-CHOP-14, R-CHOP-21) is acceptable. Liposomal doxorubicin, epirubicin, or pirarubicin (also known as therarubicin) is acceptable. R-EPOCH is acceptable.
6. Patients' last treatment with R-chemotherapy must be 6 to 14 weeks prior to start of study drug.
7. Patients with ECOG performance status (PS) 0, 1, or 2.
8. Patients willing to provide a portion of his/her tumor tissue from original diagnosis or lymph node to confirm diagnosis.
9. The following laboratory values obtained ≤ 21 days prior to start of study drug:

   * Absolute neutrophil count ≥ 1000/mm3 (or 1.0 GI/L, SI units)
   * Platelet count ≥ 100,000/mm3 (or 100 GI/L, SI units)
   * Hemoglobin ≥ 9 g/dL (can be achieved by transfusion)
   * Total bilirubin ≤ 2 x ULN (if >2 x ULN direct bilirubin is required and should be ≤1.5 x ULN)
   * AST ≤ 3 x ULN
   * Serum creatinine ≤ 2 x ULN
10. Women of childbearing potential must have had a negative serum pregnancy test 14 days prior to the start of study drug plus a negative local urine pregnancy test on Day 1, Cycle 1 prior to treatment and must be willing to use adequate methods of contraception during the study and for 8 weeks after study drug administration.
11. Patients who give a written informed consent obtained according to local guidelines.
12. Patients capable of swallowing intact study medication tablets and following directions regarding taking study drug, or have a daily caregiver who will be responsible for administering study drug.

Exclusion Criteria:

1. Patients with evidence of disease according to the revised IWRC (Cheson et al 2007) after completion of the first-line R-chemotherapy treatment, prior to study entry.
2. Patients receiving ongoing radiation therapy or who received radiation therapy to the residual tumor masses < 4 weeks from start of study drug.
3. Patients who have previously received systemic mTOR inhibitor (sirolimus, temsirolimus, everolimus, etc).
4. Patients with evidence of current central nervous system (CNS) involvement with lymphoma. Patients who have only had prophylactic intrathecal chemotherapy against CNS disease are eligible.
5. Patients with transformed follicular lymphoma.
6. Patients who received ibritumomab tiuxetan (Zevalin®), in order to avoid potential delayed kidney toxicities.
7. Patients who had myelosuppressive chemotherapy or biologic therapy < 3 weeks from start of study drug.
8. Patients receiving chronic systemic immunosuppressive agents. Inhaled and topical steroids are acceptable. Patients may be receiving stable (not increased within the last month) chronic doses of corticosteroids with a maximum dose of 20 mg of prednisone or ≤5 mg of dexamethasone per day, if they are being given for disorders other than lymphoma such as rheumatoid arthritis, polymyalgia rheumatica, adrenal insufficiency or asthma.
9. Patients with active, bleeding diathesis.
10. Patients with a known history of HIV seropositivity.
11. Patients with known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to any of the excipients.
12. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

    * unstable angina pectoris, symptomatic congestive heart failure (NYHA II, III, IV), myocardial infarction ≤ 6 months prior to first study drug, serious uncontrolled cardiac arrhythmia, cerebrovascular accidents ≤ 6 months before study drug start
    * severely impaired lung function as defined as spirometry and DLCO that is ≤ 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
    * poorly controlled diabetes as defined by fasting serum glucose >2.0 x ULN
    * any active (acute or chronic) or uncontrolled infection/disorders that impair the ability to evaluate the patient or for the patient to complete the study
    * nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by this study drug, such as severe hypertension that is not controlled with medical management and thyroid abnormalities whose thyroid function cannot be maintained in the normal range by medication
    * liver disease such as cirrhosis or decompensated liver disease.
13. Patients who have a history of another primary malignancy ≤ 3 years, with the exception of non-melanoma skin cancer and carcinoma in situ of uterine cervix.
14. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes.
15. Patients who are using other investigational agents or who had received investigational drugs ≤ 4 weeks prior to study drug start.
16. Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2009-07-24 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (178):
- United States (34):
  - Ironwood Cancer and Research Centers SC, Chandler, Arizona
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - University of California San Diego - Moores Cancer Center Dept of Moores Cancer Ctr (3), La Jolla, California
  - USC/Kenneth Norris Comprehensive Cancer Center Dept.ofNorrisMedicalCenter(4), Los Angeles, California
  - University of Colorado Health, Colorado Springs, Colorado
  - Denver Health & Hospital Authority CACZ885M2301, Denver, Colorado
  - Rocky Mountain Cancer Centers RMCC, Greenwood Village, Colorado
  - University Cancer Institute, Boynton Beach, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Columbus Regional, Columbus, Georgia
  - Rush University Medical Center Div. of Hematology & Oncology, Chicago, Illinois
  - Indiana University Hospital IU Cancer Center, Indianapolis, Indiana
  - Tulane University Health Sciences Center Office of Clinical Research, New Orleans, Louisiana
  - Lahey Clinic Dept of Lahey Clinic (3), Burlington, Massachusetts
  - Mayo Clinic - Rochester Dept. of MayoClinic-Rochester, Rochester, Minnesota
  - Washington University School of Medicine Div. of Medical Oncology, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center Dartmouth, Lebanon, New Hampshire
  - Levine Cancer Institute Oncology, Charlotte, North Carolina
  - Wake Forest University Baptist Medical Center Dept. of WFUHS, Winston-Salem, North Carolina
  - University of Pittsburgh Medical Center SC-3, Pittsburgh, Pennsylvania
  - Medical University of South Carolina -Hollings Cancer Center MUSC/HCC (2), Charleston, South Carolina
  - Cancer Centers of the Carolinas Cancer Centers of Carolinas (3, Greenville, South Carolina
  - University of Tennessee Cancer Institute SC-2, Memphis, Tennessee
  - The West Clinic, Memphis, Tennessee
  - The Center for Cancer and Blood Disorders Dept. of The Ctr for C & BD, Fort Worth, Texas
  - University of Texas/MD Anderson Cancer Center Dept of MD Anderson (18), Houston, Texas
  - Baylor College of Medicine Dept.of Baylor College of Med., Houston, Texas
  - South Texas Oncology and Hematology, PA South Texas Oncology (2), San Antonio, Texas
  - Texas A&M HealthSciencesCtr-Scott & White Memorial Hospital CenterForCancerPrevention&Care, Temple, Texas
  - University of Vermont Office of Clinical Trials Res., Burlington, Vermont
  - University of Virginia Health Systems SC-2, Charlottesville, Virginia
  - Blue Ridge Research Center at Roanoke Neurological Center SC, Roanoke, Virginia
  - Dean Health System, Madison, Wisconsin
  - Waukesha Memorial Hospital Cancer Center Dept.ofWaukeshaMemorialHosp., Waukesha, Wisconsin
- Argentina (3):
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Australia (4):
  - Novartis Investigative Site, Douglas, Queensland
  - Novartis Investigative Site, Greenslopes, Queensland
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Geelong, Victoria
- Austria (4):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Leoben
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Brazil (4):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (8):
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- China (5):
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Colombia (3):
  - Novartis Investigative Site, Bogotá, Cundinamarca
  - Novartis Investigative Site, Bucaramanga
  - Novartis Investigative Site, Medellín
- Czechia (4):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Olomouc, CZE
  - Novartis Investigative Site, Prague
- Egypt (3):
  - Novartis Investigative Site, Al Mansurah
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- France (6):
  - Novartis Investigative Site, Amiens Cedex1
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Saint-Priest-en-Jarez
- Germany (8):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, München
- Greece (4):
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Ioannina, GR
  - Novartis Investigative Site, Athens
- Novartis Investigative Site, Hong Kong, Hong Kong
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- Israel (5):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (18):
  - Novartis Investigative Site, Brindisi, BR
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Piacenza, PC
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Potenza, PZ
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Venezia, VE
- Japan (14):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Kure, Hiroshima
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Shinjuku-ku, Japan
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Sunto-gun, Shizuoka
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Koto, Tokyo
  - Novartis Investigative Site, Fukuoka
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, Saida
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
- New Zealand (2):
  - Novartis Investigative Site, Grafton, Auckland
  - Novartis Investigative Site, Wellington
- Novartis Investigative Site, Oslo, Norway
- Peru (2):
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
- Poland (4):
  - Novartis Investigative Site, Lublin, Lublin Voivodeship
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Warsaw
- Russia (4):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
- Saudi Arabia (3):
  - Novartis Investigative Site, Dammam
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Bratislava, Slovakia
- South Korea (2):
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Korea
- Spain (12):
  - Novartis Investigative Site, Cadiz, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Zurich, CH
  - Novartis Investigative Site, Bellinzona
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Songkhla
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Talas / Kayseri
- Novartis Investigative Site, Caracas, Distrito Federal, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Witzig TE, Tobinai K, Rigacci L, Ikeda T, Vanazzi A, Hino M, Shi Y, Mayer J, Costa LJ, Bermudez Silva CD, Zhu J, Belada D, Bouabdallah K, Kattan JG, Kuruvilla J, Kim WS, Larouche JF, Ogura M, Ozcan M, Fayad L, Wu C, Fan J, Louveau AL, Voi M, Cavalli F. Adjuvant everolimus in high-risk diffuse large B-cell lymphoma: final results from the PILLAR-2 randomized phase III trial. Ann Oncol. 2018 Mar 1;29(3):707-714. doi: 10.1093/annonc/mdx764. PMID 29253068
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/webapp/etrials/searchTrial.do?t=i&trialID=755&keywords=crad001n2301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Considering a recruitment period of 53 months and a final primary analysis performed after an anticipated duration of 69 months after study start, 727 patients had to be included. Actual enrolled: 742.
Groups:
- RAD001 (Everolimus)1: RAD001 10 mg (two 5 mg tablets), daily for 12 months
- Placebo: Everolimus placebo 10 mg (two 5 mg tablets), daily for 12 months
Period: Overall Study
Arm/Group | RAD001 (Everolimus)1 | Placebo
Started | 372 | 370
Untreated Participants | 4 (not treated due to administrative problems, protocol deviation, and subject withdrawal of consent.) | 6 (not treated due to administrative problems and subject withdrawal of consent.)
Completed | 177 (completed = treatment duration completed as per protocol) | 249 (completed = treatment duration completed as per protocol)
Not Completed | 195 | 121
Not completed — Abnormal lab values | 3 | 2
Not completed — Administrative problems | 5 | 9
Not completed — Adverse Event | 113 | 44
Not completed — Death | 1 | 0
Not completed — Disease progression | 24 | 48
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 10 | 2
Not completed — Withdrawal by Subject | 18 | 7
Not completed — Subject/guardian decision | 20 | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) includes all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | RAD001 (Everolimus)1 | Placebo | Total
Number analyzed (Participants) | 372 | 370 | 742
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (13.72) | 60.9 (13.61) | 60.7 (13.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 166 | 370
  Male | 168 | 204 | 372

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: DFS was defined as the time from date of randomization to the date of event defined as the first documented relapse of the disease or death due to any cause. Relapse was based on investigator assessment and was assigned only if: It was documented according to Cheson guidelines by an objective radiological assessment method; It was documented by a biopsy proven lymphoma including new or recurrent bone marrow involvement; A new anticancer therapy for lymphoma started with subsequent confirmation of the relapse within 4 weeks of the start of this anticancer therapy
Time Frame: From date of randomization to the date of event defined as the first documented recurrence of the disease, or death due to any cause and up to 6 years
Population: Full Analysis Set (FAS) includes all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RAD001 (Everolimus)1 | Placebo
Number analyzed (Participants) | 372 | 370
Percentage of participants | 77.8 [72.7 to 82.1] | 77.0 [72.1 to 81.1]
Statistical Analysis 1: Comparison: RAD001 (Everolimus)1 vs Placebo; Test type: Superiority or Other; p = 0.276, Log Rank — P-value was obtained from the one-sided unstratified log rank test; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.69 to 1.22]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to date of death due to any cause. If the patient was not known to have died, survival was censored at the date of the last contact.
Time Frame: From date of randomization to date of death due to any cause up to around 7 years
Population: Full Analysis Set (FAS) includes all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RAD001 (Everolimus)1 | Placebo
Number analyzed (Participants) | 372 | 370
Percentage of participants
  2 years | 90.7 [87.0 to 93.4] | 88.3 [84.4 to 91.3]
  3 years | 88.0 [83.8 to 91.1] | 83.7 [79.3 to 87.3]
  4 years | 85.4 [80.7 to 89.1] | 80.7 [75.8 to 84.7]
  5 years | 83.4 [78.1 to 87.5] | 77.4 [71.7 to 82.0]
  6 years | 80.3 [71.6 to 86.6] | 77.4 [71.7 to 82.0]
Statistical Analysis 1: Comparison: RAD001 (Everolimus)1 vs Placebo; Test type: Superiority or Other; There was no formal testing of the OS between treatment since the primary endpoint was not statistically significant; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.52 to 1.09]

3. Secondary Outcome: Lymphoma-specific Survival (LSS)
Description: LSS was defined as time from randomization to death as a result of lymphoma.
Time Frame: From randomization to death documented as a result of lymphoma up to 7 years
Population: Full Analysis Set (FAS) includes all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RAD001 (Everolimus)1 | Placebo
Number analyzed (Participants) | 372 | 370
Percentage of participants
  2 years | 94.9 [91.8 to 96.8] | 90.5 [86.9 to 93.2]
  3 years | 93.1 [89.6 to 95.5] | 88.8 [84.9 to 91.8]
  4 years | 91.6 [87.6 to 94.3] | 86.9 [82.6 to 90.3]
  5 years | 89.4 [84.6 to 92.8] | 85.4 [80.5 to 89.2]
  6 years | 89.4 [84.6 to 92.8] | 85.4 [80.5 to 89.2]
Statistical Analysis 1: Comparison: RAD001 (Everolimus)1 vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.41 to 1.07]

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Groups:
- RAD001 (Everolimus): RAD001 10 mg (two 5 mg tablets), daily for 12 months
- All Patients: All Patients in the Everolimus and Placebo groups.
Arm/Group | RAD001 (Everolimus) | Placebo | All Patients
Serious Adverse Events (participants affected / at risk) | 105/368 | 62/364 | 167/732
Other Adverse Events (participants affected / at risk) | 348/368 | 276/364 | 624/732
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (Everolimus) (N=368) | Placebo (N=364) | All Patients (N=732)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 3
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 5 | 13
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 7 | 4 | 11
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 3
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 3
Atrial flutter (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 4 | 2 | 6
Cardiac failure congestive (Cardiac disorders) | 5 | 1 | 6
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 1 | 2
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0 | 2
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 1
Cataract (Eye disorders) | 1 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 1
Ophthalmoplegia (Eye disorders) | 0 | 1 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 1
Vision blurred (Eye disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2
Disease progression (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 2 | 0 | 2
Pyrexia (General disorders) | 3 | 2 | 5
Sudden death (General disorders) | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1 | 3
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 1 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 2
Cellulitis (Infections and infestations) | 2 | 1 | 3
Cytomegalovirus colitis (Infections and infestations) | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 1
Enteritis infectious (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 1 | 3
Hepatitis B (Infections and infestations) | 1 | 2 | 3
Herpes zoster (Infections and infestations) | 1 | 1 | 2
Implant site infection (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 1
Moraxella infection (Infections and infestations) | 1 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 | 1 | 4
Pneumonia (Infections and infestations) | 7 | 3 | 10
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 1
Pneumonia cryptococcal (Infections and infestations) | 1 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 1
Pyonephrosis (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 2 | 0 | 2
Skin infection (Infections and infestations) | 0 | 1 | 1
Systemic infection (Infections and infestations) | 0 | 1 | 1
Tinea pedis (Infections and infestations) | 0 | 1 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 3 | 4
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Biopsy lung (Investigations) | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 2 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 3
Lymphocyte count decreased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Brachial plexopathy (Nervous system disorders) | 0 | 1 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Encephalomalacia (Nervous system disorders) | 0 | 1 | 1
Facial paresis (Nervous system disorders) | 0 | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
IVth nerve paresis (Nervous system disorders) | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1
Optic neuritis (Nervous system disorders) | 0 | 1 | 1
Paraparesis (Nervous system disorders) | 0 | 2 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 1 | 1
Vocal cord paresis (Nervous system disorders) | 0 | 1 | 1
Device difficult to use (Product Issues) | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 3
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1
Testicular swelling (Reproductive system and breast disorders) | 0 | 1 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Granulomatous pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Arteriosclerosis (Vascular disorders) | 0 | 2 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 2
Erythromelalgia (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 1 | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0 | 1
Varicose ulceration (Vascular disorders) | 1 | 0 | 1
Vein disorder (Vascular disorders) | 1 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (Everolimus) (N=368) | Placebo (N=364) | All Patients (N=732)
Anaemia (Blood and lymphatic system disorders) | 61 | 18 | 79
Leukopenia (Blood and lymphatic system disorders) | 29 | 23 | 52
Lymphopenia (Blood and lymphatic system disorders) | 22 | 13 | 35
Neutropenia (Blood and lymphatic system disorders) | 89 | 57 | 146
Thrombocytopenia (Blood and lymphatic system disorders) | 55 | 9 | 64
Abdominal pain (Gastrointestinal disorders) | 25 | 21 | 46
Aphthous ulcer (Gastrointestinal disorders) | 21 | 4 | 25
Constipation (Gastrointestinal disorders) | 19 | 25 | 44
Diarrhoea (Gastrointestinal disorders) | 99 | 49 | 148
Dry mouth (Gastrointestinal disorders) | 23 | 5 | 28
Mouth ulceration (Gastrointestinal disorders) | 57 | 13 | 70
Nausea (Gastrointestinal disorders) | 51 | 37 | 88
Stomatitis (Gastrointestinal disorders) | 166 | 28 | 194
Vomiting (Gastrointestinal disorders) | 34 | 30 | 64
Asthenia (General disorders) | 37 | 28 | 65
Fatigue (General disorders) | 66 | 55 | 121
Oedema peripheral (General disorders) | 69 | 25 | 94
Pyrexia (General disorders) | 62 | 32 | 94
Nasopharyngitis (Infections and infestations) | 42 | 32 | 74
Pneumonia (Infections and infestations) | 23 | 3 | 26
Sinusitis (Infections and infestations) | 21 | 11 | 32
Upper respiratory tract infection (Infections and infestations) | 42 | 27 | 69
Urinary tract infection (Infections and infestations) | 20 | 18 | 38
Blood cholesterol increased (Investigations) | 21 | 5 | 26
Blood lactate dehydrogenase increased (Investigations) | 33 | 5 | 38
CD4 lymphocytes decreased (Investigations) | 37 | 18 | 55
Weight decreased (Investigations) | 28 | 6 | 34
Decreased appetite (Metabolism and nutrition disorders) | 43 | 19 | 62
Hypercholesterolaemia (Metabolism and nutrition disorders) | 42 | 13 | 55
Hyperglycaemia (Metabolism and nutrition disorders) | 40 | 26 | 66
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 32 | 16 | 48
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 31 | 61
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 33 | 55
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 28 | 53
Dizziness (Nervous system disorders) | 21 | 27 | 48
Dysgeusia (Nervous system disorders) | 25 | 7 | 32
Headache (Nervous system disorders) | 42 | 31 | 73
Insomnia (Psychiatric disorders) | 25 | 16 | 41
Cough (Respiratory, thoracic and mediastinal disorders) | 65 | 40 | 105
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 | 11 | 43
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 34 | 2 | 36
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 24 | 1 | 25
Pruritus (Skin and subcutaneous tissue disorders) | 36 | 22 | 58
Rash (Skin and subcutaneous tissue disorders) | 70 | 31 | 101
Hypertension (Vascular disorders) | 19 | 13 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.